CLINICAL TRIAL: NCT03405857
Title: Effects of the Cognitive Enhancing Information & Communication Technology (ICT) Contents in Patients With Mild Cognitive Impairment
Brief Title: Effects of the Cognitive Enhancing ICT Contents in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-01-013-010
Record Dates: First submitted 2018-01-01; First posted 2018-01-23 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2017-12

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; cognitive training program
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Cognitive rehabilitation program will be administered for 4 weeks, three times a week, 30 minutes a day
  Interventions: Other: Cognitive rehabilitation program
- Group 2 (No Intervention): No intervention will be administered

INTERVENTIONS:
Other: Cognitive rehabilitation program — Cognitive rehabilitation programs have been developed to improve the cognitive functions of the elderly or patients with cognitive impairments. The program includes sub-categories such as attention, working memory, memory and executive functions with various levels of difficulty.
  Other Names: Computer-aided Cognitive Rehabilitation Training System
  Arms: Group 1

SUMMARY:
The purpose of this study is to investigate the effect of cognitive rehabilitation program on the improvement of cognitive functions in patients with mild cognitive impairment(MCI).

DETAILED DESCRIPTION:
The cognitive rehabilitation program was developed to improve cognitive functions of the elderly or patients with cognitive impairments. The study will enroll 40 patients with mild cognitive impairment(MCI) between 55 and 75 years of age. Forty subjects will be randomly assigned into two groups. Subjects in the intervention group will receive four weeks of cognitive rehabilitation training, three times per week and 30 minutes per day. The control group will not receive any intervention. The investigator will measure their cognitive and brain functions three times at pre-intervention, post-intervention and four weeks after intervention to assess the effectiveness of the cognitive training program.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with mild cognitive impairment through clinical interview, neuropsychological tests and brain imaging
* No history of neurologic diseases

Exclusion Criteria:

* Severe cognitive problems(MMSE<10)
* Other psychiatric disorder including bipolar or schizophrenic disorder
* Other problems disturbing cognitive tests

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-04-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline performance on Digit Span Test (Neuropsychological test) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It measures auditory attention span and includes forward and backward trials. The participant listens to a series of numbers and calls the sequence correctly. The sequence increases in each trial. The final score is the longest number of sequential digits that the participant can remember correctly. The scores range from 3 to 8. The higher the score, the better the performance.
Change from baseline performance on Visual Span Test (Neuropsychological test) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It measures spatial attention span and includes forward and backward trials. The participant will see sequence of blocks "lit up" on a computer screen, and then repeat the sequence in order or back in order. The sequence increases in each trial. The final score is the longest number of sequential blocks that the participant can remember correctly. The scores range from 3 to 8. The higher the score, the better the performance.
Change from baseline performance on Visual Continuous Performance Test (Neuropsychological test) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It measures a participant's visual sustained and selective attention. The participant will see numbers from "0" to "9" presented on a computer screen and they must click the mouse when "3" appeared. The test will run for 9 minutes. The main scores produced in this test are omission errors, commission errors and reaction times. Higher score means worse performance.
Change from baseline performance on Auditory Continuous Performance Test (Neuropsychological test) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It measures a participant's auditory sustained and selective attention. The participant will hear numbers from "0" to "9", and when they hear "3" they must click the mouse. The test will run for 9 minutes. The main scores produced in this test are omission errors, commission errors and reaction times. Higher score means worse performance.
Change from baseline performance on Trail Making Test (Neuropsychological test) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It consists of type A and type B trials. The participant should connect the numbers (1~25) as quickly as possible in type A trial, and connect the numbers (1~13) and alphabets (A~L) alternatively as quickly as possible in type B trial. The main scores produced in this test are completion time and errors. Higher score means worse performance.
Change from baseline performance on Stroop test (Neuropsychological test) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It measures a participant's processing speed, selective attention and inhibitory control. The participant will be asked to read 'word' of the colored words or 'name of the color' of the colored words in separate trials. The main scores produced in this test are completion time and errors. The contrast score of the two trial's completion time means interference.
Change from baseline performance on Visual Recognition test (Neuropsychological test) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It measures participant's visual memory. The participant will see 15 visual patterns presented on a computer screen and recognize them immediately. The participant will be asked to recognize the 15 patterns after 20 minutes again. The main scores produced in this test are the numbers of recognized patterns in immediate and delayed trials. Immediate memory score is the sum of 5 trial's correct response and score ranges between 0 and 60. Delayed memory score is the correct response of the delayed trial and the score range is 0 to 15. Higher score means better performance.
Change from baseline performance on Auditory Verbal Learning test (Neuropsychological test) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It measures participant's verbal memory. The participant will hear 15 words and recall them immediately and after 20 minutes again. The main scores produced in this test are the numbers of recalled words of the immediate and delayed trials. Immediate memory score is the sum of 5 trial's correct response and score ranges between 0 and 60. Delayed memory score is the correct response of the delayed trial and the score range is 0 to 15. Higher score means better performance.

SECONDARY OUTCOMES:
Change from baseline score on Korean Version of Geriatric Depression Test Short Form (Depression scale) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It measures depressive symptoms of the participants. The score ranges between 0 and 15. Higher score means severe depression.
Change from baseline activity on functional Near-Infrared Spectroscopy (fNIRS) at 4 weeks and 8 weeks | baseline, 4 weeks and 8 weeks
  It measures brain activity during cognitive tasks to see if cognitive training affects brain function.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea